CLINICAL TRIAL: NCT00773266
Title: Intraocular Architecture of Secondary Implanted Anterior Chamber Iris-Fixated Lenses in Aphakic Eyes Evaluated With Anterior Segment Optical Coherence Tomography
Brief Title: Intraocular Position of Secondary Iris-Fixated IOLs in Aphakic Eyes
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Michael Koss, PI, Johann Wolfgang Goethe University Hospital
Other Study IDs: MK-APHAKIA-08
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Aphakia
Keywords: Aphakia; Secondary IOL-Implantation; Iris-Fixated IOL; Artisan; Anterior Segment OCT; Aphakia - secondary iris-fixated IOL position
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the intraocular stability and safety of secondary iris-fixated IOLs in aphakic patients.

DETAILED DESCRIPTION:
18 eyes of 16 patients received secondary anteriorly iris-fixated intraocular lenses (IOLs) to correct for aphakia without capsular support, partly combined with anterior or complete pars plana vitrectomy. Primary outcome measurements included visual acuity (6m Snellen charts), central endothelium cell count (cECC) and postoperative intraocular position of the IOL assessed with anterior segment optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with aphakia due to complicated cataract surgery, weakness in lens support (capsula, zonulae) Marfans´s syndrome

Exclusion Criteria:

* Aphakia due to preexisting corneal, retinal o uveal disease, low endothelial cell count

Ages: 16 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with long standing Aphakia and eligibility for secondary IOL implantantion were retrospectively examined
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Intraocular IOL position | 12-35 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für Augenheilkunde, Frankfurt am Main, Hesse, Germany